CLINICAL TRIAL: NCT02140541
Title: The Clinical Profile of UK Asthma Patients With Raised Blood Eosinophils
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Other Study IDs: R05812
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Asthma
Keywords: Asthma; Blood eosinophils; Sputum eosinophils; Clinical predictor; UK primary care; Global Initiative for Asthma (GINA)
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Blood eosinophil count ≤ 400/µl
- Blood eosinophil count > 400/µl

SUMMARY:
To explore the relationship between blood eosinophil counts, asthma exacerbations and patient asthma control using a large primary care based research database

DETAILED DESCRIPTION:
Sputum eosinophil levels have been shown to predict asthma exacerbation and inhaled corticosteroid (ICS) responsivenesss. Managing asthma based on sputum eosinophils leads to fewer exacerbations than management adhering to Global Initiative for Asthma (GINA) guidelines. However the use of sputum to measure eosinophil levels is expensive and impractical within a clinical setting. This study explores the use of blood-eosinophil levels as a clinical predictor for exacerbations and asthma control within a UK primary care dataset.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 12-80 at date of last eosinophil count
* Asthma diagnosis at any time
* Blood Eosinophil reading in patient record (numeric count expressed in µl) at least one year prior to last data extraction
* Two years of continuous data

Exclusion Criteria:

* Any other chronic respiratory diseases
* Eosinophil counts >5000/µl (outliers)

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A retrospective database analysis of asthma patients with a valid eosinophil count (where valid: numeric value expressed as /µl at least one year prior to last data extraction) with at least one year of data of prior to the date of eosinophil count (baseline period) and one year of data post recorded eosinophil count (outcome period).
Sampling Method: Non-Probability Sample
Enrollment: 130248 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Exacerbations | 1 year
  Defined as:
  * American Thoracic Society / European Respiratory Society (ATS/ERS) task force definition: Asthma related hospital admissions OR accident and emergency (A&E) room attendance OR Use of acute oral steroids
  * Clinical definition: ATS/ERS definition including any GP consultations for lower respiratory related tract infections (LRTIs) treated with antibiotics
Asthma control | 1 year
  Defined as:
  * Risk domain asthma control: No Asthma-related hospital attendance, A&E attendance, out-patient department attendance, no prescriptions for acute oral steroids and no GP consultations for LRTIs treated with antibiotics
  * Overall asthma control: Risk domain asthma control definition, including average daily dose of ≤200mcg salbutamol

CONTACTS AND LOCATIONS:
Overall Officials: David Price, Prof, MD, Principal Investigator — University of Aberdeen
Locations (1):
- Research in Real Life Ltd, Cambridge, United Kingdom

REFERENCES:
- [Background] Deykin A, Lazarus SC, Fahy JV, Wechsler ME, Boushey HA, Chinchilli VM, Craig TJ, Dimango E, Kraft M, Leone F, Lemanske RF, Martin RJ, Pesola GR, Peters SP, Sorkness CA, Szefler SJ, Israel E; Asthma Clinical Research Network, National Heart, Lung, and Blood Institute/NIH. Sputum eosinophil counts predict asthma control after discontinuation of inhaled corticosteroids. J Allergy Clin Immunol. 2005 Apr;115(4):720-7. doi: 10.1016/j.jaci.2004.12.1129. PMID 15805990
- [Background] Green RH, Brightling CE, McKenna S, Hargadon B, Parker D, Bradding P, Wardlaw AJ, Pavord ID. Asthma exacerbations and sputum eosinophil counts: a randomised controlled trial. Lancet. 2002 Nov 30;360(9347):1715-21. doi: 10.1016/S0140-6736(02)11679-5. PMID 12480423
- [Derived] Price DB, Rigazio A, Campbell JD, Bleecker ER, Corrigan CJ, Thomas M, Wenzel SE, Wilson AM, Small MB, Gopalan G, Ashton VL, Burden A, Hillyer EV, Kerkhof M, Pavord ID. Blood eosinophil count and prospective annual asthma disease burden: a UK cohort study. Lancet Respir Med. 2015 Nov;3(11):849-58. doi: 10.1016/S2213-2600(15)00367-7. Epub 2015 Oct 19. PMID 26493938